CLINICAL TRIAL: NCT05919069
Title: A Single Dose, Non-Randomised, Open-Label, Parallel Group Study to Investigate the Effect of Hepatic Impairment on the Pharmacokinetics, Safety and Tolerability of AZD2693
Brief Title: A Phase I Study to Investigate the Effect of Hepatic Impairment on the PK, Safety, and Tolerability of AZD2693
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: D7830C00008
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Hepatic Impairment
Keywords: Mild; Moderate; Severe; Healthy Matches
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled within the following groups based on their CP classification score as determined at screening: Group 1: Participants with mild hepatic impairment (CP Class A, score of 5 or 6).
  Group 2: Participants with moderate hepatic impairment (CP Class B, score of 7 to 9).
  Group 3: Participants with severe hepatic impairment (CP Class C, score of 10 to 15).
  Group 4: Participants with normal hepatic function matched on a group level regarding age, body weight, and sex to the impaired groups
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Participants with mild hepatic impairment (CP Class A, score of 5 or 6)
  Interventions: Drug: AZD2693
- Group 2 (Experimental): Participants with moderate hepatic impairment (CP Class B, score of 7 to 9)
  Interventions: Drug: AZD2693
- Group 3 (Experimental): Participants with severe hepatic impairment (CP Class C, score of 10 to 15)
  Interventions: Drug: AZD2693
- Group 4 (Experimental): Participants with normal hepatic function matched on a group level regarding age, body weight, and sex to the impaired groups
  Interventions: Drug: AZD2693

INTERVENTIONS:
Drug: AZD2693 — Subcutaneous administration of AZD2693 single dose in participants with hepatic impairment

SUMMARY:
Subcutaneous administration of AZD2693 single dose in participants with hepatic impairment

DETAILED DESCRIPTION:
This is a Phase I, multicentre, single-dose, non-randomised, open-label, parallel-group study to examine the PK, safety, and tolerability of AZD2693 administered as an subcutaneous injection in male and female participants with mild, moderate, or severe hepatic impairment compared with male and female participants with normal hepatic function (as control). Eight participants with mild impairment (CP Class A); 8 participants with moderate impairment (CP Class B); 8 participants with severe impairment (CP Class C); and 8 to12 participants with normal hepatic function matched on a group level regarding age, body weight, and sex to the impaired participants are planned for study intervention with the goal of having at least 6 evaluable participants within each group. Study participants who self-withdraw after study intervention may be replaced to ensure that at least 6 participants per group are evaluable and complete the study per protocol. An evaluable participant is defined as having adequate plasma PK profile to meet the primary study objective. Child-Pugh scoring, detailed in Table 2, will be used to determine the level of hepatic impairment. Participants will be enrolled into the following groups based on their CP classification score as determined at screening: Group 1: Participants with mild hepatic impairment (CP Class A, score of 5 or 6).

Group 2: Participants with moderate hepatic impairment (CP Class B, score of 7 to 9).

Group 3: Participants with severe hepatic impairment (CP Class C, score of 10 to 15).

Group 4: Participants with normal hepatic function.

Study Arms and Duration:

* Planned screening duration per participant: up to 4 weeks.
* Planned study duration (screening to follow-up) per participant: up to 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

For Hepatic:

* Participant with a diagnosis of chronic and stable hepatic impairment

For Healthy:

* Participant with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or 12-lead ECGs,

All participants:

- Body weight ≥ 50 kg; BMI within the range of 18.0 to 40.0 kg/m2 (inclusive) as measured at screening

Exclusion Criteria:

* Participant with impaired hepatic function has eGFR < 60 mL/minute/1.73 m2 and participant with normal hepatic function has eGFR < 90 mL/minute/1.73 m2
* Positive test for HIV at screening
* History or presence of clinically significant thyroid disease
* History or presence of clinically significant or unstable medical or psychiatric condition
* History of any major surgical procedure within 30 days prior to study intervention

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
PK parameters AUCinf | 85 days
  area under the concentration-time curve (AUC) from zero to infinity (AUCinf)
PK parameters AUClast | 85 days
  area under the concentration-time curve from time zero to last time of quantifiable concentration
PK parameters Cmax | 85 days
  maximum observed plasma concentration

SECONDARY OUTCOMES:
PK parameters tmax | 85 days
  tmax: time to maximum observed plasma concentration
PK parameters tlast | 85 days
  tlast: time of the last measurable concentration
PK parameters t1/2λz | 85 days
  apparent terminal elimination half-life
PK parameters CL/F | 85 days
  CL/F: apparent clearance
PK Parameters Vz/F | 85 days
  Vz/F: apparent volume of distribution based on terminal phase
PK parameters CLR | 85 days
  CLR: Renal clearance of drug from plasma
PK parameters fe | 85 days
  fe: Percentage of dose excreted unchanged in urine
PK parameters Ae | 85 days
  Amount of unchanged drug excreted into urine

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Research Site, Rialto, California
  - Research Site, Miami Lakes, Florida
  - Research Site, Orlando, Florida